CLINICAL TRIAL: NCT05370261
Title: Comparing the Pharmacological Profile of Different Berberine Formulations, and Their Effects on Blood Sugar Levels
Brief Title: Pharmacological Profile of Different Berberine Formulations, and Effects on Blood Sugar Levels
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Factors Group of Nutritional Companies Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2021-08-004
Record Dates: First submitted 2022-05-04; First posted 2022-05-11 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Pharmacokinetics
Keywords: Bioavailability; Berberine; LipoMicel; Pharmacokinetics

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Berberine LipoMicel soft-gel (Experimental): Each participant receives their treatment of Berberine LipoMicel soft-gel capsules at a total dose of 500 mg berberine. Treatments are consumed with a glass of water (approx. 200 mL), and standardized breakfast. A standardized lunch is served after the 4hr fasting; standardized dinner after 8hrs. Capillary whole blood samples are collected at time points 0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24 hours.
  Samples that are not processed the same day are kept frozen at -20°C until further processing and analysis. Processed samples are analyzed by LC-MS within 24 hours after processing.
  Participants are asked to arrive after an overnight fast (at least 9hrs). Each participant acts as their own control; there is no separate control group. A washout period of at least 7 days between each treatment will be used.
  Adverse events are recorded throughout the study by direct questioning.
  Interventions: Dietary Supplement: Berberine LipoMicel
- Regular Berberine hard-gel (Experimental): Each participant receives their treatment of regular Berberine hard-gel capsules at a total dose of 500 mg berberine. Treatments are consumed with a glass of water (approx. 200 mL), and standardized breakfast. A standardized lunch is served after the 4hr fasting; standardized dinner after 8hrs. Capillary whole blood samples are collected at time points 0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24 hours.
  Samples that are not processed the same day are kept frozen at -20°C until further processing and analysis. Processed samples are analyzed by LC-MS within 24 hours after processing.
  Participants are asked to arrive after an overnight fast (at least 9hrs). Each participant acts as their own control; there is no separate control group. A washout period of at least 7 days between each treatment will be used.
  Adverse events are recorded throughout the study by direct questioning.
  Interventions: Dietary Supplement: Regular Berberine hard-gels

INTERVENTIONS:
Dietary Supplement: Berberine LipoMicel — Berberine LipoMicel® soft-gels. Total dose of 500 mg of berberine
  Arms: Berberine LipoMicel soft-gel
Dietary Supplement: Regular Berberine hard-gels — Total dose of 500 mg of berberine
  Arms: Regular Berberine hard-gel

SUMMARY:
The primary objective of this study is to evaluate the gastrointestinal absorption of berberine (hydrochloride) in a novel formulation in healthy adult volunteers by comparing it with free berberine (hydrochloride) formulation. Several pharmacokinetic parameters are compared.

As secondary objective, the immediate or short-term effects of Berberine supplementation on blood sugar levels in healthy volunteers are evaluated via a glucose tolerance test (OGTT) using a portable glucometer.

ELIGIBILITY:
Inclusion Criteria:

* Age 21-65
* healthy, good physical condition

Exclusion Criteria:

* Pregnancy or breast-feeding
* Gastrointestinal conditions
* Acute or chronic liver disease
* Acute or chronic kidney disease
* Acute or chronic cardiovascular disease
* Hematological disease
* Diabetes
* Allergy or Intolerance to gluten
* Allergy or Intolerance to Berberine
* Use of any form of nicotine or tobacco
* Alcohol and substance abuse history
* Use of medications (e.g., blood sugar-lowering agents, or statins)
* Use of Berberine supplements
* Participation in another investigational study

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-05-04 (Actual); Study Completion 2022-05-04 (Actual)

PRIMARY OUTCOMES:
AUC: the area under the concentration-time curve | 0 (baseline; pre-dose), 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24 hours (post-dose)
  To evaluate the gastrointestinal absorption of orally ingested berberine (hydrochloride) in a novel formulation in healthy adult volunteers by comparing the Area under the plasma concentration versus time curve (AUC) with that of with free/regular berberine (hydrochloride).
Cmax: maximum plasma concentration | 0 (baseline; pre-dose), 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24 hours (post-dose)
  To evaluate the gastrointestinal absorption of orally ingested berberine (hydrochloride) in a novel formulation in healthy adult volunteers by comparing the Peak Plasma Concentration (Cmax) with that of with free/regular berberine (hydrochloride).
Tmax: the time point of maximum plasma concentration | 0 (baseline; pre-dose), 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24 hours (post-dose)
  To evaluate the gastrointestinal absorption of orally ingested berberine (hydrochloride) in a novel formulation in healthy adult volunteers by comparing the time point of maximum plasma concentration (Tmax) with that of with free/regular berberine (hydrochloride).

SECONDARY OUTCOMES:
Effects on Blood sugar levels | 0 (Baseline; pre-dose), 0.5, 1, 2, 3, and 4 hours (post-dose)
  To evaluate the immediate or short-term effects of orally ingested Berberine on blood sugar levels in healthy volunteers by using a glucose tolerance test (OGTT).
Changes in Blood sugar concentrations | 0 (Baseline; pre-dose), 0.5, 1, 2, 3, and 4 hours (post-dose)
  To evaluate changes in blood sugar concentrations of orally ingested Berberine in healthy volunteers by using a portable glucometer.

CONTACTS AND LOCATIONS:
Locations (1):
- ISURA, Burnaby, British Columbia, Canada

REFERENCES:
- [Derived] Solnier J, Zhang Y, Kuo YC, Du M, Roh K, Gahler R, Wood S, Chang C. Characterization and Pharmacokinetic Assessment of a New Berberine Formulation with Enhanced Absorption In Vitro and in Human Volunteers. Pharmaceutics. 2023 Nov 1;15(11):2567. doi: 10.3390/pharmaceutics15112567. PMID 38004546